CLINICAL TRIAL: NCT03890627
Title: Interest of Cardiac Output Measurement by Thoracic Bio-reactance for Monitoring of Patients Treated for a Pulmonary Hypertension
Brief Title: Thoracic Bio-reactance Measurement of Cardiac Output in Pulmonary Hypertension
Acronym: PHREACT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0819
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic bio-reactance measurement of cardiac output
  Interventions: Device: Thoracic bio-reactance

INTERVENTIONS:
Device: Thoracic bio-reactance — Cardiac output variation measured by thoracic bio-reactance, between inclusion and one year after hemodynamic evaluation by right cardiac catheterization, to discriminate stable patients from those that degrade.

SUMMARY:
Pulmonary Hypertension (PH) is a rare disease characterized by an increase in pulmonary vascular resistance, leading to a progressive decline in cardiac output (CO).Since cardiac output is correlated with the prognosis of the disease, the conduct of a right heart catheterization (thermodilution measurement, reference technique) during the annual follow-up visit of patients in competences centres is recommended. In practice, it is not systematically performed because of it is invasive, with potential risk for the patient, and there is limited logistical capacity for its implementation. The estimation of cardiac output is thus often based on cardiac ultrasound but its measurement is potentially biased.

Starling ™ SV is a non-invasive cardiac output monitor based on thoracic bio-reactance measurement. Several clinical studies have shown that cardiac output measured by bio-reactance is strongly correlated with the measurement obtained by catheterization in different indications. Rich et al. (2013) assessed bio-reactance specifically in 50 patients with Pulmonary Hypertension compared with thermodilution. The results showed that the measurement of cardiac output by bio-reactance was feasible in these patients, had a better accuracy than by catheterization, and was reliable for detecting changes in cardiac output after a vasodilatation test.

The Starling ™ SV monitor could thus have a place in the follow-up of patients who are being treated for Pulmonary Hypertension. Since it is a rapid, non-invasive examination, it could be performed on an outpatient basis, especially as a first-line test to check the stability of the CO, thus avoiding the systematic use of right heart catheterization, which would then be reserved only to patients for whom the measurement by bio-reactance would show a decrease of cardiac output compared to the previous value. Before being able to propose this use in current practice, it is necessary to carry out a pilot study which will make it possible to explore the interest of bio-reactance in this situation.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Presenting pulmonary hypertension (PH) followed by the Competence Center of the Hospices Civils de Lyon
* Follow-up for pulmonary hypertension groups 1, 4 or 5
* Of which the cardiac index is ≥ 2,5 L/min/m²
* Expressing its non-opposition to the participation of this study
* Benefiting from a social security scheme or similar

Exclusion Criteria:

* Adult patient protected by Law
* Patient for whom a thermodilution measurement of cardiac output (CO) is unreliable: right-left shunt; or uncorrected congenital heart disease; or variability> 10% of the 3 measurements of CO obtained by thermodilution
* pulmonary hypertension groups 2 or 3
* Hemodynamic aggravation since the previous visit: increased pressure or decreased cardiac index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pulmonary hypertension and followed by a Competence Center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Ability of the relative variation of cardiac output measured by thoracic bio-reactance to predict the patient's status (stable or unstable). | 12 months
  A patient will be considered unstable if the decrease in the relative variation of cardiac output measured with thermodilution between visit one and one year after visit one is at least 15%. Then, the ability of the relative variation of cardiac output measured by thoracic bio-reactance to predict the patient's status (stable or unstable) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Explorations Fonctionnelles Respiratoires, centre de compétences de l'hypertension pulmonaire Hospices Civils de Lyon, Groupement Hospitalier Est, Bron, France

IPD SHARING:
Plan to Share IPD: No